CLINICAL TRIAL: NCT05276609
Title: ARTEMIS-001: A Phase 1, Open-label, Multi-center Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of Multiple Doses of Intravenous Administration of HS-20093 in Patients With Locally Advanced or Metastatic Solid Tumors Who Have Progressed Following Prior Therapy
Brief Title: ARTEMIS-001: Phase 1 Study of the HS-20093 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Hansoh Biomedical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Hansoh BioMedical R&D Company (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-20093-101
Record Dates: First submitted 2022-02-18; First posted 2022-03-11 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced solid tumor; B7-H3; antibody-drug conjugate (ADC); HS-20093

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-20093 (Phase Ia: Dose escalation) (Experimental): There are seven escalating dose cohorts.
  Interventions: Drug: HS-20093 (Phase Ia: Dose escalation)
- HS-20093 (Phase Ib: Dose expansion) (Experimental): The recommended dose from the dose-escalation stage and other potential doses will be further explored.
  Interventions: Drug: HS-20093 (Phase Ib: Dose expansion)

INTERVENTIONS:
Drug: HS-20093 (Phase Ia: Dose escalation) — Intravenous (IV) administration of HS-20093 Q3W; Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.
  Arms: HS-20093 (Phase Ia: Dose escalation)
Drug: HS-20093 (Phase Ib: Dose expansion) — IV administration of HS-20093 Q3W; Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.
  Arms: HS-20093 (Phase Ib: Dose expansion)

SUMMARY:
HS-20093 is a fully humanized IgG1 antibody-drug conjugate (ADC) which specifically binds to B7-H3, a target wildly expressed on solid tumor cells. The objectives of this study are to investigate the safety, tolerability, pharmacokinetics and anti-tumor activity of HS-20093 in Chinese advanced solid tumor patients.

This is a phase 1, open-label, multi-center, dose-escalation and expansion study evaluating the safety, tolerability, pharmacokinetic (PK), and the therapeutic potential of HS-20093 as a monotherapy in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multi-center, dose-escalation and expansion, first-in-human phase 1 study in Chinese adult participants with locally advanced or metastatic solid tumors. This study will consist of two parts: A Part Ia dose escalation stage and a Part Ib dose expansion stage.

The objectives of this study are to evaluate the safety, tolerability, PK and preliminary anti-tumor activity, describe the dose-limiting toxicities (DLTs), and determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) of HS-20093.

Part Ia: Participants with advanced cancer are eligible for dose escalation study if they have progressed on or intolerant to available standard therapies, or no standard or available curative therapy exists. The dose escalation will include an initial accelerated titration design followed by i3+3 design.

Part Ib: Enrollment into dose expansion will begin after identification of the MTD or MAD in Phase Ia. The dose expansion study will be conducted in populations with the following indications: locally advanced or metastatic non- small cell lung cancer (NSCLC)，extensive stage small cell lung cancer (ES-SCLC) and other types of advanced solid tumor.

All patients will be carefully followed for adverse events during the study treatment and for 90 days after the last dose of study drug. Subjects will be permitted to continue therapy with assessments for progression if the product is well tolerated and sustained clinical benefit exists.

ELIGIBILITY:
Inclusion Criteria:

1. At least age of 18 years at screening;
2. Histologically or cytologically confirmed, locally advanced or metastatic solid tumors for which standard treatment either does not exist or has proven ineffective or unavailable or intolerable
3. At least one extra-cranial measurable lesion according to RECIST 1
4. Agree to provide fresh or archival tumor tissue
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0~1
6. Life expectancy >= 12 weeks
7. Agree to use medically accepted methods of contraception
8. Men or women should be using adequate contraceptive measures throughout the study;
9. Females subjects must not be pregnant at screening or have evidence of non-childbearing potential
10. Signed and dated Informed Consent Form

Exclusion Criteria:

Any of the following would exclude the subject from participation in the study:

1. Treatment with any of the following:

   * Previous or current treatment with B7-H3 targeted therapy
   * Any cytotoxic chemotherapy, investigational agents and anticancer drugs within 14 days prior to the first scheduled dose of HS-20093
   * Prior treatment with a monoclonal antibody within 28 days prior to the first scheduled dose of HS-20093
   * Radiotherapy with a limited field of radiation for palliation within 2 weeks, or patients received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks prior to the first scheduled dose of HS-20093
   * Major surgery within 4 weeks prior to the first scheduled dose of HS-20093
2. Subjects with previous or concurrent malignancies
3. Inadequate bone marrow reserve or organ dysfunction
4. Evidence of cardiovascular risk
5. Evidence of current severe or uncontrolled systemic diseases
6. Evidence of mucosal or internal bleeding within 1 month prior to the first scheduled dose of HS-20093
7. Known active infection requiring antibodies treatment within 2 weeks, or severe infection within 4 weeks prior to the first scheduled dose of HS-20093
8. Subjects with current infectious diseases
9. History of neuropathy or mental disorders
10. Pregnant or lactating female
11. History of severe hypersensitivity reaction, severe infusion reaction or idiosyncrasy to drugs chemically related to HS-20093 or any of the components of HS-20093
12. Known vaccination or hypersensitivity of any level within 4 weeks prior to the first scheduled dose of HS-20093
13. Unlikely to comply with study procedures, restrictions, and requirements in the opinion of the investigator
14. Any disease or condition that, in the opinion of the investigator, would compromise subject safety or interfere with study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2021-11-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Ⅰa (Dose-Escalation Stage): Maximum tolerated dose (MTD) for HS-20093 | Up to day 21 from the first dose
  To determine the MTD for further evaluation of IV administration of HS-20093 in subjects with advanced solid tumors.
Ⅰb (Dose-Expansion Stage): Objective response rate (ORR) determined by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | From the first dose up to PD or withdrawal from study, whichever came first, assessed up to 24 months
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). ORR is evaluated by the number of participants with best overall response of complete response (CR) and partial response (PR) [Confirmed CR/PR assessment require at least one repeat (≥4 weeks)].

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From the first dose through 90 days post end of treatment
  AE assessed by investigator exclusively related to subject's underlying disease or medical condition [graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0]. Any untoward medical occurrence in a clinical study participant, whether or not considered related to the medicinal product. Incidence and severity of AEs are assessed according to vital signs, laboratory variables, physical examination, electrocardiogram, etc.
Observed maximum plasma concentration (Cmax) of HS-20093 in participants with advanced solid tumor | From pre-dose to 14 days after the first dose on Cycle 1
  Cmax will be obtained following administration of the first dose of HS-20093 during the first cycle.
Time to reach maximum plasma concentration (Tmax) of HS-20093 following the first dose in participants with advanced solid tumor | From pre-dose to 14 days after the first dose on Cycle 1
  Tmax will be obtained following administration of the first dose of HS-20093 during the first cycle.
Terminal half-life (T1/2) of HS-20093 following IV dose in participants with advanced solid tumor | From pre-dose to 14 days after the first dose on Cycle 1
  Apparent terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz.
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) following the first dose of HS-20093 | From pre-dose to 14 days after the first dose on Cycle 1
  Area under the plasma concentration versus time curve from time zero to the last sampling time when the concentration was no less than the lower limit of quantification (LLQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
Percentage of participants with antibodies to HS-20093 in serum | From pre-dose to 90 days post end of treatment
  Serum samples were collected for the determination of anti-drug antibody (ADA) at designated time points.
ORR determined by investigators according to RECIST 1.1 (dose-escalation stage) | From the first dose up to PD or withdrawal from study, whichever came first, assessed up to 24 months
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). ORR is evaluated by the number of participants with best overall response of CR and PR (Confirmed CR/PR assessment require at least 1 repeat).
Duration of response (DOR) determined by investigators according to RECIST 1.1 | From the first dose up to PD or death, whichever came first, assessed up to 24 months
  DoR was defined as the period from the first occurrence of CR or PR to PD or death from any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) would be used [Confirmed CR/PR assessment require at least one repeat (≥4 weeks)].
Disease control rate (DCR) determined by investigators according to RECIST 1.1 | From the first dose up to PD or withdrawal from study, whichever came first, assessed up to 24 months
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). DCR was evaluated by the number of participants with best overall response of CR, PR and stable disease (SD) [Confirmed CR/PR assessment require at least one repeat (≥4 weeks); SD shall be assessed at least 5 weeks after the first dose].
Progression-free survival (PFS) determined by investigators according to RECIST 1.1 | From the randomization/first dose up to PD or death, whichever came first, assessed up to 24 months
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). PFS was defined as the time from random assignment (dose expansion stage) or first dose (dose escalation stage) to PD or death from any cause.
Overall survival (OS) (only in dose expansion stage) | From the randomization/first dose up to death, whichever came first, assessed up to 24 months
  OS was defined as the time from random assignment (dose expansion stage) or first dose (dose escalation stage) to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No